CLINICAL TRIAL: NCT00280527
Title: Protocol for the Assessment of Variability in Histology and Gene Expression in Bariatric Surgery Patients.
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary Rinella, Mary E. Rinella, MD, Northwestern University, Northwestern University
Other Study IDs: 1347-004
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Obesity
Keywords: NAFLD; NASH; Obesity; Bariatric Surgery; Weight Reduction
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Weight Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is known that a vast majority of patients seeking a bariatric surgery weight reduction procedure have non-alcoholic fatty liver disease (NAFLD), while a smaller subset of patients within this group have a more serious liver problem known as nonalcoholic steatohepatitis (NASH). NASH is a serious liver disease that can lead to cirrhosis, liver failure and ultimately liver transplantation. The purpose of this study is to explore the effects of bariatric surgery on the progression of NASH. The investigators also hope to gain insight into which genes may be responsible for the development of NAFLD and NASH. The knowledge gained from this study will advance the field of fatty liver disease and help design rational treatments to prevent disease progression.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of abnormal liver tests in the United States. NAFLD is often found in association with obesity and diabetes and it is expected to become increasingly prevalent as the incidence of diabetes and obesity continues to increase. NAFLD represents a range of diseases from simple fatty deposition in the liver to more aggressive inflammation and fibrosis, termed nonalcoholic steatohepatitis (NASH). The distinction of NASH as an entity within NAFLD is an important one, as the natural history of this disease is different. Ultimately, NASH may progress to cirrhosis in up to 25% of patients, compared to simple steatosis which is a benign condition.

NAFLD has been estimated at 10-24% in various populations and is significantly higher in obese populations (57.5-74%). NASH is a subset of NAFLD characterized by fatty change with lobular inflammation, hepatocellular injury, progressive fibrosis and cirrhosis. The bariatric surgery population is an ideal cohort to study a large subset of NASH; those with morbid obesity.

The purpose of this study is to examine variability of hepatic histology as well as expression of key metabolic genes in NAFLD/NASH patients undergoing bariatric surgery. Patients will undergo pre-operative laboratory testing, followed by intra-operative liver and fat biopsies. A 12-month follow up will consist of repeat liver biopsy and laboratory testing. We predict that histologic variability of inflammation and fibrosis in NASH is accompanied by differential gene expression. Furthermore, if this variability is pronounced, this will temper the reliance on percutaneous liver biopsy in NASH as the "gold standard" and further emphasize the need for global markers of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to give written informed consent
* Subjects must fulfill the criteria for bariatric surgery that have been recommended by a National Institutes of Health (NIH) consensus conference.

These criteria include:

1. The patient should be greater than 100 pounds above desirable body weight or a Body Mass Index (BMI) >40 kg/m2.
2. Presence of significant obesity-related illnesses with a BMI of 35-40 kg/m2.
3. Failure of sustained weight loss on supervised dietary and/or medical regimens.
4. Patient shows understanding of the risks and benefits of surgery and understands lifestyle changes subsequent to the operation.
5. Acceptable operative risk.

   * Adult subjects 18-65 years of age of any race or gender

Exclusion Criteria:

* Anti - smooth muscle Ab < 1:80.
* Serum Hepatitis B surface antigen (HepBsAg) negative.
* Serum Hepatitis C Antibody (HepC Ab) negative
* Iron/TIBC ratio (transferrin saturation) < 45%
* Alpha-1-antitrypsin level within normal limits
* Ceruloplasmin level within normal limits.
* Negative pregnancy test (females)
* No active drug abuse or within 6 months
* Etoh consumption < 20g/day (males) or < 10 g/day (females) - Assessed by one physician and confirmed with one family member.
* No known diagnosis of malignancy
* Any other conditions which the investigator feels would make the subject unsuitable for enrollment, or could interfere with the subject completing the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective trial of obese patients with presumed NAFLD undergoing bariatric surgery. Patients will be enrolled at Northwestern Memorial Hospital through the bariatric surgery clinic.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2006-09; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Rinella, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States